CLINICAL TRIAL: NCT01014169
Title: A Randomized Controlled Trial of The Impact of Parental Note Taking on the Effectiveness of Anticipatory Guidance: the Suzuki Music Model Applied to Urban Pediatrics
Brief Title: Study of the Impact of Parental Note Taking on the Effectiveness of Anticipatory Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: The Joel and Barbara Alpert Endowment For The Children of The City (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-28356
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-09

CONDITIONS: Health Education; Sudden Infant Death
Keywords: Health education; Sudden Infant Death; Breast Feeding; Infant Equipment
MeSH Terms: conditions — Health Education; Sudden Infant Death; Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Mothers in the control group will receive the nursing discharge newborn information from the nurse practitioner [sometimes via a Spanish interpreter, if required] according to current standard of care, which includes verbal information and written handouts.
- Note taking (Experimental): The mothers in the intervention group will be given a pen and encouraged to take written notes in the notes section of the discharge envelope using their language of preference when receiving the standard newborn information.
  Interventions: Behavioral: Note taking

INTERVENTIONS:
Behavioral: Note taking — The mothers in the intervention group will be given a pen and encouraged to take written notes in the notes section of a discharge envelope using their language of preference when receiving standard newborn discharge information.
  Arms: Note taking

SUMMARY:
The delivery of anticipatory guidance is an essential component of pediatric practice. Given the large amount of information to be shared during each encounter and the limited time available, there is a need for an effective and efficient means of communication between health care providers and families. The investigators hypothesize that more active parental participation in the form of note taking during the delivery of anticipatory guidance will lead to increased knowledge, higher levels of satisfaction with the encounter, and increased adoption of recommended parenting practices.

In this study, the investigators propose a randomized controlled trial of the impact of note taking during the delivery of newborn anticipatory guidance on maternal practices related to newborn care. The investigators plan to compare a control group of mothers receiving standard of care anticipatory guidance with an intervention group of mothers who are encouraged to take written notes while receiving the anticipatory guidance. The primary outcome of interest is maternal practice related to infant sleep position, and the secondary outcomes of interest are maternal practice related to breastfeeding initiation and car seat use. The investigators also plan to evaluate the impact of note taking on mothers' knowledge of recommended practices related to newborn care and on mothers' satisfaction with the guidance received.

DETAILED DESCRIPTION:
The importance of communicating effectively with families and children is not unique to medicine. In the field of child music education, research has shown that effective parental involvement is linked to musical achievement [1]. The Suzuki method of music education in particular emphasizes this involvement and regards an effective teacher-child-parent relationship as fundamental to learning [2]. Parental engagement both during the music lesion and at home is key, and parents are routinely encouraged to take notes during the lesson so they can accurately recall the instruction for practice at home [1]. The Suzuki method is based on the idea that this model of education can be used with any family in any environment [3]. We are interested to learn whether a similar approach can be applied to pediatric anticipatory guidance in an urban population.

Note taking has been shown to improve both memory and comprehension in a number of settings. In a study of memory aids, participants taking notes exhibited higher levels of accurate recall of information than participants using other techniques [4]. Another study demonstrated that participants who took notes and then had the notes to review had improved recall of information when compared to participants who were given written information to study but did not take notes themselves [5]. Even doodling has been shown to lead to improved memory and to aid with concentration [6]. Interestingly, patient or family note taking for retention of medical information has not been extensively studied.

A number of studies have been done to look at interventions to improve both the delivery of health information and the retention of the information provided. Randomized controlled trials have looked at the impact of specific training programs for providers [7] and at practice-wide changes in office systems [8], and have shown improvements in the amount and quality of guidance provided. A study looking at the impact of physician advice on behavior change found that patients who had received counseling by their physician prior to receiving related written materials had better recall of information and were more likely to share the materials with others when compared to patients who only received the written material with no counseling [9]. A study on information recall of instructions given in the emergency department for otitis media care showed that parents retained more information at one and three days after the encounter when they received either standardized verbal or written instructions, as opposed to the usual verbal instructions [10].

The effective delivery of health information plays a central role in pediatric primary care. In 1990, the Federal Maternal and Child Health Bureau, along with the American Academy of Pediatrics, launched Bright Futures, a set of health supervision guidelines for pediatric patients aged birth to 21 [11]. The guidelines, which provide a framework for well-patient care, emphasize a partnership between the healthcare team, the family, and the child and highlight a number of recommended topics to be covered at routine visits [12]. This is a standard curriculum for primary care in many pediatric residencies, including the Boston Combined Residency Program.

For many families, the first interaction with a healthcare provider for their child occurs during the newborn evaluation prior to discharge from the hospital. The newborn anticipatory guidance recommended by Bright Futures is divided into the five categories of family readiness, infant behaviors, feeding, safety, and routine newborn care [12]. Included in these topics are recommendations for counseling on prone sleeping position, or "back to sleep," breast feeding support, and car seat use, all of which have been shown to improve infant health and safety [13,14,15]. Despite the recommendations for newborn anticipatory guidance, a national survey of parents with young children showed that 38% of parents reported never having discussed newborn care with a healthcare provider [16]. The authors of the study comment that it is difficult to know whether a portion of these families received information but were unable to remember it at the time of the survey. In the same study, a perceived lack of information was correlated with decreased satisfaction with care. The parents who reported discussing fewer anticipatory guidance topics gave their providers lower overall ratings.

A survey of sleep position of infants seen at an urban primary care center in Washington DC showed that 34.1% of infants were sleeping in the recommended supine position [17]. A subsequent study of sleep position reported by parents of black infants at a WIC clinic in Washington DC showed that 57.7% of the infants were sleeping in the supine position [13]. While there are many factors that impact parental behaviors around sleep position, the most common reasons given for supine sleeping position in this study were concern for SIDS and advice from a health care professional. These findings indicate that improved delivery of anticipatory guidance may play a role in increasing the proportion of infants sleeping on their backs.

At Boston Medical Center (BMC), a group of three nurse practitioners split full-time coverage of the newborn nursery and are responsible for doing a great deal of the newborn teaching with parents. Prior to discharge from the hospital, each infant is evaluated and teaching on newborn care is done using both verbal instruction and written handouts. This teaching, which is based on the Bright Futures recommendations, covers topics including feeding, diaper care, bathing, dressing, umbilical cord care, circumcision care, safety, sleeping, and crying. The providers also review warning signs that may indicate that an infant is sick. At the time this teaching is done, each mother is given a large envelope containing the discharge documents. On the outside of the envelope is a section designated for taking notes, although this is not currently used by the providers or parents.

In our study, a randomized controlled trial, we will draw on the techniques promoted by the Suzuki method of music education to see if the principles of increased parental involvement and parental note taking can improve information retention and impact behavior change. We hypothesize that more active parental participation in the form of note taking during the delivery of anticipatory guidance will lead to increased knowledge, higher levels of satisfaction with the encounter, and increased adoption of recommended parenting practices. Our specific aims are as follows:

Specific Aim 1: To evaluate the impact of note taking during the delivery of newborn anticipatory guidance on maternal behavior. The primary outcome of interest is maternal practice related to infant sleep position, and the secondary outcomes of interest are maternal practice related to breastfeeding initiation and car seat use.

Specific Aim 2: To evaluate the impact of note taking on mothers' knowledge of recommended practices related to newborn care.

Specific Aim 3: To evaluate the impact of note taking during health information delivery on mothers' satisfaction with the guidance received.

ELIGIBILITY:
Inclusion Criteria:

* newborn gestational age greater than 35 weeks
* maternal spoken fluency in either English or Spanish
* a working telephone in the home.

Exclusion Criteria:

* either the newborn or the mother has a medical condition requiring hospitalization for longer than 4 days after a cesarean section or 2 days after a vaginal delivery
* mother not expected to retain custody of the infant at the time of discharge

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Jason Wang, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kendall J. Suzuki's Mother Tongue Method. Music Educators Journal. 1986;72:47-50
- [Background] Creech A and Hallam S. Parent-teacher-pupil interactions in instrumental music tuition: a literature review. B.J. Music Ed. 2003;20:29-44.
- [Background] Grilli S. An interview with Dr. Shin'ichi Suzuki at the Talent Education Institute. International Review of Education. 1992; 38: 547-551.
- [Background] Intons-Peterson MJ, Fournier J. External and Internal Memory Aids: When and How Often Do We Use Them? Journal of Experimental Psychology: General. 1986;115:267-280.
- [Background] Kiewra KA DuBois NF, McShane CD, et al. Note-taking functions and techniques. Journal of Educational Psychology. 1991;83:240-245.
- [Background] Andrade J. What Does Doodling Do? Appl Cognit Psychol.2009;23:1-7.
- [Background] Gielen AC, Wilson ME, McDonald EM, Serwint JR, Andrews JS, Hwang WT, Wang MC. Randomized trial of enhanced anticipatory guidance for injury prevention. Arch Pediatr Adolesc Med. 2001 Jan;155(1):42-9. doi: 10.1001/archpedi.155.1.42. PMID 11177061
- [Background] Rosenthal MS, Lannon CM, Stuart JM, Brown L, Miller WC, Margolis PA. A randomized trial of practice-based education to improve delivery systems for anticipatory guidance. Arch Pediatr Adolesc Med. 2005 May;159(5):456-63. doi: 10.1001/archpedi.159.5.456. PMID 15867120
- [Background] Kreuter MW, Chheda SG, Bull FC. How does physician advice influence patient behavior? Evidence for a priming effect. Arch Fam Med. 2000 May;9(5):426-33. doi: 10.1001/archfami.9.5.426. PMID 10810947
- [Background] Isaacman DJ, Purvis K, Gyuro J, Anderson Y, Smith D. Standardized instructions: do they improve communication of discharge information from the emergency department? Pediatrics. 1992 Jun;89(6 Pt 2):1204-8. PMID 1594378
- [Background] Green M, Kessel SS. Diagnosing and treating health: bright futures. Pediatrics. 1993 May;91(5):998-1000. No abstract available. PMID 8474827
- [Background] 2008. Bright Futures: Guidelines for Health Supervision of Infants, Children, and Adolescents, Third Edition. Elk Grove Village, IL: American Academy of Pediatrics.
- [Background] Moon RY, Oden RP, Grady KC. Back to Sleep: an educational intervention with women, infants, and children program clients. Pediatrics. 2004 Mar;113(3 Pt 1):542-7. doi: 10.1542/peds.113.3.542. PMID 14993547
- [Background] United States Preventative Services Task Force: Recommendations of Breastfeeding Counseling. www.ahrq.gov/clinic/uspstf/uspsbrfd.htm. Accessed on 11/25/08.
- [Background] Zaza S, Sleet DA, Thompson RS, Sosin DM, Bolen JC; Task Force on Community Preventive Services. Reviews of evidence regarding interventions to increase use of child safety seats. Am J Prev Med. 2001 Nov;21(4 Suppl):31-47. doi: 10.1016/s0749-3797(01)00377-4. PMID 11691560
- [Background] Schuster MA, Duan N, Regalado M, Klein DJ. Anticipatory guidance: what information do parents receive? What information do they want? Arch Pediatr Adolesc Med. 2000 Dec;154(12):1191-8. doi: 10.1001/archpedi.154.12.1191. PMID 11115301
- [Background] Moon RY, Omron R. Determinants of infant sleep position in an urban population. Clin Pediatr (Phila). 2002 Oct;41(8):569-73. doi: 10.1177/000992280204100803. PMID 12403373

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mothers on the postpartum ward of an urban safety-net hospital were recruited. Inclusion criteria included gestational age > 35 weeks, fluency in English or Spanish, and access to a telephone. Mothers were excluded if there was prolonged hospitalization of the mother or the infant or if they were not expected to retain custody of the infant.
Groups:
- Usual Care: Mothers in the control group received newborn information from the nurse practitioner [sometimes via a Spanish interpreter, if required] according to current standard of care, which includes verbal information and written handouts.
- Note Taking: The mothers in the intervention group were given a pen and paper and encouraged to take written notes using their language of preference when receiving the standard newborn information.
Period: Overall Study
Arm/Group | Usual Care | Note Taking
Started | 65 | 61
Completed | 58 | 48
Not Completed | 7 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Note Taking | Total
Number analyzed (Participants) | 65 | 61 | 126
Age Continuous [Mean (Standard Deviation); unit: years] | 27.8 (6.5) | 28.9 (6.4) | 28.3 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 61 | 126
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 32 | 63
  Not Hispanic or Latino | 34 | 29 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 20 | 42
  White | 7 | 9 | 16
  More than one race | 30 | 30 | 60
  Unknown or Not Reported | 0 | 0 | 0
Language [Number; unit: participants]
  English | 37 | 36 | 73
  Spanish | 28 | 25 | 53
Number of pregnancies [Median (Inter-Quartile Range); unit: Pregnancies] | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]
Number of Children [Median (Inter-Quartile Range); unit: Children] | 2 [2 to 2] | 2 [1 to 2] | 2 [2 to 2]
Type of delivery [Number; unit: participants]
  Vaginal | 46 | 46 | 92
  Cesarean section | 19 | 15 | 34
Type of Insurance [Number; unit: participants]
  Medicaid | 52 | 46 | 98
  Free Care | 5 | 3 | 8
  Private | 7 | 11 | 18
  None | 1 | 1 | 2
Highest Education Level [Number; unit: participants]
  Less than/some high school | 24 | 14 | 38
  High school graduate | 15 | 21 | 36
  Vocational/trade school | 1 | 2 | 3
  Some college | 9 | 11 | 20
  Associates degree | 5 | 1 | 6
  Bachelors degree | 7 | 7 | 14
  Graduate/professional degree | 4 | 5 | 9
Received prenatal care [Number; unit: participants]
  Yes | 65 | 61 | 126
  No | 0 | 0 | 0
Attended Childbirth Classes [Number; unit: participants]
  Yes | 10 | 12 | 22
  No | 55 | 49 | 104
Other Adults in the Home [Number; unit: participants]
  No other adult in home | 9 | 8 | 17
  Spouse/partner | 43 | 44 | 87
  Baby's grandmother | 10 | 12 | 22
  Baby's grandfather | 6 | 4 | 10
  Baby's uncles or aunts | 17 | 11 | 28
  Other adult | 2 | 2 | 4
Nurse Practitioner [Number; unit: participants]
  Patients Seen By Nurse Practitioner # 1 | 37 | 34 | 71
  Patients Seen By Nurse Practitioner # 2 | 21 | 22 | 43
  Patients Seen By Nurse Practitioner # 3 | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome of Interest is Maternal Practice Related to Supine Infant Sleep Position.
Description: This measure assesses maternal report of placing the infant on the back to sleep (supine sleep position) as opposed to putting the infant on its side or stomach.
Time Frame: two days after discharge
Measure: Number; unit: participants who report supine position
Arm/Group | Usual Care | Note Taking
Number analyzed (Participants) | 58 | 48
participants who report supine position | 45 | 42
Statistical Analysis 1: Comparison: Usual Care vs Note Taking; Test type: Superiority or Other; Risk Ratio (RR) = 1.13, 95% CI 2-sided [0.95 to 1.34]

2. Secondary Outcome: Maternal Practice Related to Breastfeeding Initiation
Description: This measure assesses maternal report of breastfeeding. The number analyzed is the number who reported any breastfeeding.
Time Frame: two days after discharge
Measure: Number; unit: participants who report breastfeeding
Arm/Group | Usual Care | Note Taking
Number analyzed (Participants) | 58 | 48
participants who report breastfeeding | 50 | 46
Statistical Analysis 1: Comparison: Usual Care vs Note Taking; Test type: Superiority or Other; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.99 to 1.25]

3. Secondary Outcome: Maternal Practice Related to Correct Car Seat Use
Description: Correct car seat use by all subjects who use cars was defined as placing the car seat in the back seat facing backwards and using the car seat every time the infant travels by car. The number reported is the number who report using the car seat correctly.
Time Frame: two days after discharge
Measure: Number; unit: participants with correct car seat use
Arm/Group | Usual Care | Note Taking
Number analyzed (Participants) | 55 | 46
participants with correct car seat use | 48 | 46
Statistical Analysis 1: Comparison: Usual Care vs Note Taking; Test type: Superiority or Other; Risk Ratio (RR) = 1.12, 95% CI [1.00 to 1.25]

ADVERSE EVENTS:
Arm/Group | Usual Care | Note Taking
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/61
Other Adverse Events (participants affected / at risk) | 0/65 | 0/61

LIMITATIONS AND CAVEATS:
Conducted as a pilot study and not powered to demonstrate a significant difference between the two groups; subjects and NPs were aware of the group assignment; outcomes were determined using maternal self report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No